CLINICAL TRIAL: NCT01878279
Title: Longitudinal Study to Evaluate the Frequency of HSV-1 Oral Reactivation in Children in Dar es Salaam, Tanzania
Brief Title: HSV Oral Reactivation in Children
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 21397
Record Dates: First submitted 2013-06-11; First posted 2013-06-14 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-06

CONDITIONS: HSV-1; HIV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV negative
- HIV positive: HIV positive children in care
  Interventions: Other: Underlying medical illness

INTERVENTIONS:
Other: Underlying medical illness
  Groups: HIV positive

SUMMARY:
In the proposed study, the investigators will carry out novel research to evaluate both symptomatic and asymptomatic daily oral herpes simplex virus (HSV) shedding rates and copy number in children with and without HIV.

Study Objectives:

1. To evaluate the frequency of oral HSV reactivation in HIV-infected and uninfected children

   Secondary Objectives:
2. To determine the acceptability of performing daily oral swabs in children age 3-12

ELIGIBILITY:
Inclusion Criteria:

* age > 3 and ≤12 years old
* parental/guardian consent and children's assent must be obtained and participants and parent/guardian must be able to comply with study procedures
* For HIV-infected group: Positive HIV serology by either ELISA x 2, ELISA + WB or PCR testing

Exclusion Criteria:

* age <3 and > 12 years old
* Acute illness which by opinion of the investigator makes enrollment in the trial unfeasible (including active tuberculosis, malaria or other opportunistic infection requiring treatment)
* co-enrollment in other therapeutic/intervention trials (observational trial enrollment is permitted).
* Stable co-administration of other medications is permitted (e.g. bactrim)
* For HIV-infected children; receiving or eligible for antiretroviral (ART) therapy by local standards

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: For this Pilot study, we will enroll 20 HIV-infected and 10 HIV-uninfected children
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-09; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
HSV detection rate | 14 days

SECONDARY OUTCOMES:
HSV copy number | 14 days

OTHER OUTCOMES:
compliance with daily swabs | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard Zuckerman, MD, MPH, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- MUHAS, Dar es Salaam, Tanzania

REFERENCES:
- [Background] Kasubi MJ, Nilsen A, Marsden HS, Bergstrom T, Langeland N, Haarr L. Prevalence of antibodies against herpes simplex virus types 1 and 2 in children and young people in an urban region in Tanzania. J Clin Microbiol. 2006 Aug;44(8):2801-7. doi: 10.1128/JCM.00180-06. PMID 16891495
- [Background] Grando LJ, Machado DC, Spitzer S, Nachman S, Ferguson F, Berentsen B, Yurgel LS. Viral coinfection in the oral cavity of HIV-infected children: relation among HIV viral load, CD4+ T lymphocyte count and detection of EBV, CMV and HSV. Braz Oral Res. 2005 Jul-Sep;19(3):228-34. doi: 10.1590/s1806-83242005000300013. Epub 2005 Nov 21. PMID 16308613